CLINICAL TRIAL: NCT04839614
Title: Concurrent Laparoscopic Hysterectomy and Weight Loss Surgery in Obese Patients With Endometrial Carcinoma or Endometrial Intraepithelial Neoplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Colleen Feltmate, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-419; NCT04278183 (obsolete NCT alias)
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Carcinoma; Obesity; EIN; Endometrial Intraepithelial Neoplasia; Endometrial Cancer Stage I
Keywords: Endometrial Carcinoma; Obesity; EIN; Endometrial Intraepithelial Neoplasia; Endometrial Cancer Stage I; Weight Loss Surgery; Bariatric Surgery
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CONCURRENT LAPAROSCOPIC HYSTERECTOMY AND WEIGHT LOSS SURGERY (Experimental): Upon enrollment in the study at first appointment with gynecologic oncologist, referral to the BWH Center for Metabolic and Bariatric Surgery (CMBS).
  * Schedule a series of appointments with a bariatric surgeon, nutritionist and psychologist, which is part of the approval process for weight loss surgery.
  * Hysterectomy and weight loss surgery will then be scheduled on the same day within 8 weeks from first visit with the gynecologic oncologist for endometrial cancer or 12 weeks if you have endometrial pre-cancer.
  * Series of post-operative visits with the bariatric surgeon and gynecologic oncologic surgeon as well as the nutritionist and psychologist.
  Interventions: Other: CONCURRENT LAPAROSCOPIC HYSTERECTOMY AND WEIGHT LOSS SURGERY-Referral

INTERVENTIONS:
Other: CONCURRENT LAPAROSCOPIC HYSTERECTOMY AND WEIGHT LOSS SURGERY-Referral — See arm description

SUMMARY:
To assess the feasibility of an expedited referral process for the obese endometrial cancer or EIN patient from her gynecologic oncologist to the Brigham Center for Metabolic and Bariatric Surgery (CMBS) in order to undergo concurrent weight loss surgery and hysterectomy within 8 weeks of first appointment with a gynecologic oncologist (or 12 weeks for EIN patients).

DETAILED DESCRIPTION:
The most common risk factor for endometrial cancer is obesity. However, because early-stage endometrial cancer has a very high survival rate, patients more often suffer from long-term issues related to their weight, like heart disease, stroke, and diabetes. Weight loss surgery has been shown to help patients lose weight and also decrease their risk for obesity-related diseases.

This research study is a Feasibility Study. This is the first-time investigators are studying both 1) the referral process of patients with endometrial cancer to the Center for Metabolic and Bariatric Surgery without delaying curative treatment of endometrial cancer 2) the combined surgery of both hysterectomy and weight loss surgery. The combined surgery of hysterectomy and weight loss surgery has been performed both at this institution and others without increased complications, but it has not been formally studied.

Approximately 30 patients are expected to participate in this study at Brigham and Women's Hospital (BWH).

ELIGIBILITY:
Inclusion Criteria:

* Female adults at least 18 years of age
* A BMI of 35-39.99 and 1 or more severe obesity-related co-morbidities

  --including T2D,112 hypertension, hyperlipidemia, obstructive sleep apnea (OSA), obesity-hypoventilation syndrome (OHS), Pickwickian syndrome (a combination of OSA and OHS), nonalcoholic 4 fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH), pseudotumor cerebri, gastroesophageal reflux disease (GERD), asthma, venous stasis disease, severe urinary incontinence, debilitating arthritis, or considerably impaired quality of life) OR a BMI ≥ 40
* Tissue diagnosis (usually endometrial biopsy) of grade 1 endometrial carcinoma or EIN.

Exclusion Criteria:

* Younger than 18 years old
* BMI < 35
* Without a tissue diagnosis, or with a grade 2 or greater endometrial cancer tissue diagnosis
* Pregnant participants will be excluded from this study.
* Patients with contraindications to bariatric surgery will also be excluded.

  --This includes active smokers, prior bariatric surgery, active substance abuse, recent suicide attempt, bulimia nervosa, large abdominal hernias, or poorly controlled psychiatric illness
* include inability to read an English informed consent form, and unwillingness to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
proportion of patients who schedule an appointment and speak with a surgeon 1-2 weeks after enrollment | 2 Weeks
  50% of the patients utilize the referral system and attend an initial consultation, it will be considered feasible
proportion of patients who undergo the concurrent surgeries within 8 weeks of diagnosis (12 weeks for EIN patients) | up 12 weeks
  concurrent surgery will be considered feasible if 50% (7-8 patients) of patients who undergo an initial consultation at the CMBS actually undergo concurrent surgery within 8 weeks of diagnosis (or 12 weeks for EIN).

SECONDARY OUTCOMES:
Safety of the concurrent surgeries | 3 weeks
  compare our safety outcomes with national complication rates for each individual surgery to assess the safety of the patient population
Postoperative complications | 3 weeks
  compare our safety outcomes with national complication rates for each individual surgery to assess the safety of the patient population
Time under anesthesia | 1 Day
  compare our safety outcomes with national complication rates for each individual surgery to assess the safety of the patient population
Total time in operating room | 1 Day
  compare our safety outcomes with national complication rates for each individual surgery to assess the safety of the patient population
Postoperative weight loss | 6 months, 1 year
  Paired t-test or Wilcoxon rank sum test will be used to compare pre- and post-surgical outcomes and survey responses
Changes in lab values reflecting comorbid conditions | 6 months, 1 year
  Paired t-test or Wilcoxon rank sum test will be used to compare pre- and post-surgical outcomes and survey responses
Post Operative 12-item Short Form Healthy Survey (SF-12) Survey | 6 months
  12-item Short Form Healthy Survey (SF-12) Survey

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Feltmate, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation